CLINICAL TRIAL: NCT06581653
Title: Medication Adherence to Phone-supervised Pancreatic Enzyme Replacement Therapy，a Prospective Randomized Clinical Trial
Brief Title: Medication Adherence to Phone-supervised Pancreatic Enzyme Replacement Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MAPPER
Record Dates: First submitted 2024-08-18; First posted 2024-09-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pancreatitis; Pancreatic Exocrine Insufficiency
Keywords: Chronic Pancreatitis; Pancreatic exocrine insufficiency; Pancreatic Enzyme Replacement Therapy; Medication Adherence
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEI Intervention Group (Experimental): 1. After enrollment, a fecal elastase-1 (FE-1) test will be conducted. If the FE-1 level is below 200ug/g, the patient will undergo a comprehensive 20-minute "WWH" medication health education session and complete a 2-week medication health assessment.
  2. Following enrollment, patients will receive monthly regular telephone counseling sessions (total of 6) to monitor medication adherence, as well as a follow-up visit at 6 months. Additionally, the MMAS-8 score for medication adherence and SF36 score for quality of life will be assessed. Patients attending the follow-up visit will undergo PEI testing using the PEI test kit. For those unable to attend in person for any reason, PEI assessment can be completed by mailing in specimens.
  3. After enrolling for 6 months, routine counseling services will cease and a follow-up visit at 12 months will take place. The MA score at 12 months will be recorded while observing the clinical course of the disease.
  Interventions: Behavioral: Phone-based PERT education intervention
- PEI Control group (No Intervention): 1. After enrollment, a fecal elastase-1 (FE-1) test will be conducted. If the FE-1 level is below 200ug/g, the patient will undergo a comprehensive 20-minute "WWH" medication health education session and complete a 2-week medication health assessment.
  2. After enrollment, patients were not frequently communicated by phone to supervise their medication, and were followed up once at the 6th and 12th month (2 times in total).Additionally, the MMAS-8 score for medication adherence and SF36 score for quality of life will be assessed.
- non-PEI Intervention Group (Experimental): 1. After enrollment, a fecal elastase-1 (FE-1) test will be conducted. If the FE-1 level is ≥ 200ug/g, the patient will undergo a comprehensive 20-minute "WWH" medication health education session and complete a 2-week medication health assessment.
  2. Following enrollment, patients will receive monthly regular telephone counseling sessions (total of 6) to monitor medication adherence, as well as a follow-up visit at 6 months. Additionally, the MMAS-8 score for medication adherence and SF36 score for quality of life will be assessed. Patients attending the follow-up visit will undergo PEI testing using the PEI test kit. For those unable to attend in person for any reason, PEI assessment can be completed by mailing in specimens.
  3. After enrolling for 6 months, routine counseling services will cease and a follow-up visit at 12 months will take place. The MA score at 12 months will be recorded while observing the clinical course of the disease.
  Interventions: Behavioral: Phone-based PERT education intervention
- non-PEI Control group (No Intervention): 1. After enrollment, a fecal elastase-1 (FE-1) test will be conducted. If the FE-1 level is ≥ 200ug/g, the patient will undergo a comprehensive 20-minute "WWH" medication health education session and complete a 2-week medication health assessment.
  2. After enrollment, patients were not frequently communicated by phone to supervise their medication, and were followed up once at the 6th and 12th month (2 times in total).Additionally, the MMAS-8 score for medication adherence and SF36 score for quality of life will be assessed.

INTERVENTIONS:
Behavioral: Phone-based PERT education intervention — Participants who allocate to the intervention group will receive regular phone-based PERT education intervention by professional team.
  Arms: PEI Intervention Group; non-PEI Intervention Group

SUMMARY:
This study aims to explore whether regular telephone intervention in patients with chronic pancreatitis can improve their Pancreatic Enzyme Replacement Therapy's Medication Adherence.

DETAILED DESCRIPTION:
Pancreatic exocrine insufficiency (PEI) represents a significant complication in cases of chronic pancreatitis (CP), exerting considerable influence on patient quality-of-life outcomes. The latest iteration (2020) from ACG's guidelines emphasizes Pancreatic Enzyme Replacement Therapy (PERT) as pivotal in managing both symptomatic and asymptomatic cases among individuals with CP. PERT not only extends median survival but also substantially mitigates symptoms while averting digestive complications associated with malabsorption-ultimately enhancing overall well-being.

An analysis revealed varying levels of PERT compliance across different patient groups-48% for those with CP, 52% for pancreatic cancer sufferers, and another 52% following pancreatic resection-induced PEI-with these rates declining to approximately 20% within one year post-initiation. Furthermore, findings from a limited-scale survey involving 148 individuals demonstrated that merely half exhibited satisfactory medication adherence; notably attributed to inadequate comprehension regarding prescribed regimens.

Presently lacking are established protocols aimed at bolstering PERT medication adherence specifically tailored towards individuals affected by CP-a gap this investigation seeks to address through comprehensive educational initiatives coupled with sustained telephonic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in the Department of gastroenterology who met the clinical diagnostic criteria of chronic pancreatitis in the 2002 Asia-Pacific Consensus Opinion in Changhai Hospital;
* at least 18 years of age;
* Have a mobile phone that can talk;
* Agree to complete the supervision and follow-up of pancreatic enzyme administration set up in this study through telephone communication.

Exclusion Criteria:

* Refusing to participate in the study;
* Exclusion of difficult differential diagnosis: diagnosis of pancreatic cancer, groove pancreatitis, and autoimmune pancreatitis within 2 years after diagnosis of chronic pancreatitis;
* Pregnant or lactating women;
* communication difficulties, mental and mental illness can not cooperate;
* There are other reasons that researchers believe should not be included (Alzheimer's disease, end-stage cancer, HIV, end-stage congestive heart failure, end-stage chronic obstructive pulmonary disease, decompensated cirrhosis, renal failure, etc.);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
MA good rate at 6 months | 6th months
  At the 6th month, the proportion of patients with good drug compliance (MMAS≥6) was in this group，The medication adherence MMAS-8 score was used, with a minimum score of 0 and a maximum score of 8, with a score of < 6 indicating poor adherence

SECONDARY OUTCOMES:
MA good rate at 12 months | 12th months
  At the 12th month, the proportion of patients with good drug compliance (MMAS≥6) was in this group,The medication adherence MMAS-8 score was used, with a minimum score of 0 and a maximum score of 8, with a score of < 6 indicating poor adherence
MA score at 6 months | 6th months
  MMAS scores of patients at the sixth month,The medication adherence MMAS-8 score was used, with a minimum score of 0 and a maximum score of 8, with a score of < 6 indicating poor adherence
MA score at 12 months | 12th months
  MMAS scores of patients aAt the 12th month,The medication adherence MMAS-8 score was used, with a minimum score of 0 and a maximum score of 8, with a score of < 6 indicating poor adherence

OTHER OUTCOMES:
Nutritional status of the patient | Average 1 year
  This data is mainly used for descriptive analysis,Height, weight, fat-soluble vitamins，The patient's height changes，weight changes by taking the drug，
Internal and external pancreatic secretory function | Average 1 year
  Exocrine function of patients Pancreatic exocrine function was assessed by fecal elastinase-1, and pancreatic endocrine function was assessed by fasting blood glucose, C-peptide,This data is mainly used for descriptive analysis,
Other adverse events associated with chronic pancreatitis in patients with chronic pancreatitis at 12 months of enrollment | Average 1 year
  The incidence of abdominal pain (frequency of attacks, VAS score), pancreatic duct stones, pancreatic pseudocyst, bile duct stenosis, cancer, severe acute pancreatitis, This data is mainly used for descriptive analysis,
Quality of Life score SF-36 | Average 1 year
  The SF-36 Quality of Life Assessment Scale quantifies a respondent's quality of life through a range of questions, including health, energy, social functioning, emotional functioning, and mental health，Based on the overall score, there are five categories: excellent (100-85), good (84-70), average (69-60), below average (59-40) and poor (≤39).

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hostipal, Shanghai, Shanghai Municipality, China